CLINICAL TRIAL: NCT04768790
Title: Effects of Multimodal Exercises Integrated With Cognitive-behavioral Therapy in Subjects With Chronic Neck Pain: a Randomized Controlled Study With One Year Follow-up
Brief Title: Effects of Multimodal Exercises Integrated With Cognitive-behavioral Therapy in Subjects With Chronic Neck Pain
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Marco Monticone, Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG/2020/16818
Record Dates: First submitted 2020-12-13; First posted 2021-02-24 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary Group (Experimental): Description of the interventions of the multidisciplinary program: multimodal exercises to improve, through gradual exposure, cervical mobility, postural control and strengthening of the cervical muscles; stabilization techniques for the deep neck muscles; task-oriented exercises maintaining the activation of the deep spinal muscle. Under the supervision of a psychologist, the subjects will also be involved in cognitive-behavioral therapy aimed at modifying the fear of movement (kinesiophobia) and the maladaptive behavior of the disease. Ergonomic consultancy.
  Interventions: Other: multidisciplinary program
- General Group (Active Comparator): Description of the interventions of the general program: exercises for muscle strengthening, regional stretching and spinal mobilization. Ergonomic consultancy.
  Interventions: Other: General program

INTERVENTIONS:
Other: multidisciplinary program — multimodal exercises to improve, through gradual exposure, cervical mobility, postural control and strengthening of the cervical muscles; stabilization techniques for the deep neck muscles; task-oriented exercises maintaining the activation of the deep spinal muscle. Under the supervision of a psychologist, the subjects will also be involved in cognitive-behavioral therapy aimed at modifying the fear of movement (kinesiophobia) and the maladaptive behavior of the disease. Ergonomic consultancy.
  Arms: Multidisciplinary Group
Other: General program — exercises for muscle strengthening, regional stretching and spinal mobilization. Ergonomic consultancy.
  Arms: General Group

SUMMARY:
The etiology of cervical pain is multifactorial and studies based on the bio-psychosocial model also link chronic neck pain to psychological factors. Among them, kinesiophobia has been reported as an important determinant. Over time, the use of multidisciplinary interventions for chronic vertebral pain (instead of segmental treatments) has grown in order to improve disability, pain and proactive behaviors towards the problem manifested. To date, the evidence relating to the effects of multidisciplinary approaches is inconclusive and lacking. In light of these premises, it appears necessary to deepen the conduct of studies aimed at evaluating the efficacy of a multidisciplinary rehabilitation program that integrates cognitive-behavioral therapy based on kinesiophobia with specific exercises, in the treatment of chronic neck pain of working subjects.

DETAILED DESCRIPTION:
Background The etiology of cervical pain is multifactorial and includes age, gender, incongruous postures, repeated efforts. Studies based on the bio-psychosocial model also link chronic neck pain to psychological factors. Among them, kinesiophobia has been reported as an important determinant. It is debatable whether interventions targeting cognitive processes and pain-associated behaviors can lead to clinically significant changes in terms of disability, pain and quality of life of these individuals.

Furthermore, there is uncertainty about the effectiveness of the types of exercises to be proposed. This makes it difficult to choose between general exercises (aimed at improving cervical muscle and joint skills) and motor-oriented (or task-oriented) exercises (aimed at cervical functional recovery in an ecological context). Over time, the use of multidisciplinary interventions for chronic vertebral pain (instead of segmental treatments) has grown in order to improve disability, pain and proactive behaviors towards the problem manifested. To date, the evidence relating to the effects of multidisciplinary approaches is inconclusive and lacking. In light of these premises, it appears necessary to deepen the conduct of studies aimed at evaluating the efficacy of a multidisciplinary rehabilitation program that integrates cognitive-behavioral therapy based on kinesiophobia with specific exercises, in the treatment of chronic neck pain of working subjects.

Hypothesis The hypothesis is that a multidisciplinary rehabilitation program induces clinically significant and long-term improvements in the disability, pain and quality of life of working subjects with chronic neck pain.

Objectives of the study Verify the effectiveness of a multidisciplinary program in inducing clinically significant and long-term improvements in the disability, pain and quality of life of working subjects suffering from chronic neck pain. Evaluate the work discomfort linked to the condition of chronic neck pain.

Study procedure The subjects eligible for the study will be assigned to one of two treatment programs (multidisciplinary or general) using a permuted block randomization procedure.

The interventions will be offered by a psychologist and two physiotherapists of equal experience, responsible separately for the multidisciplinary and general groups. Each participant will be assessed individually by postural observation, cervical and muscle mobility examination. Based on this evaluation, the exercises will be planned and performed on a single patient. Patients assigned to the multidisciplinary team will meet with a psychologist once a week.

Description of the interventions of the multidisciplinary program: multimodal exercises to improve, through gradual exposure, cervical mobility, postural control and strengthening of the cervical muscles; stabilization techniques for the deep neck muscles; task-oriented exercises maintaining the activation of the deep spinal muscle. Under the supervision of a psychologist, the subjects will also be involved in cognitive-behavioral therapy aimed at modifying the fear of movement (kinesiophobia) and the maladaptive behavior of the disease.

Description of the interventions of the general program: exercises for muscle strengthening, regional stretching and spinal mobilization.

Description of the interventions that will be carried out on both groups: ergonomic consultancy. At the end of the treatment, patients will be asked to continue with the exercises at home. At the end of each session a control of the program performed will be conducted based on a manual that includes the complete list of exercises to be performed. Patients' GPs will be asked to avoid referrals for other visits / other treatments while the programs are running.

Type of data collected:

- Personal and anthropometric data; lifestyle habits; work, pharmacological and pathological history; levels of neck disability, kinesiophobia, catastrophism, intensity of pain, quality of life, work discomfort.

Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).

At the end of the treatment, subjects will be asked to rate the effectiveness of the treatment using a Likert Global Perceived Effect scale. Using a specific form, patients will be asked to report any symptoms they experience during the study that may require further treatment.

The end date of the follow up will be considered that of December 31, 2021.

The effects of the treatment between the two groups over time will be analyzed through the use of linear models with mixed effects for repeated measurements. The differences between the two groups relating to measures with non-normal distribution will be analyzed by Mann-Whitney U test. The null hypothesis will be rejected for p values> 0.05 (two-tailed test).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic non-specific neck pain
* documented history of pain lasting more than 3 months
* good knowledge of the Italian language
* age over 18.

Exclusion Criteria:

* acute and subacute neck pain
* cognitive impairment
* presence of specific causes of neck pain (history of spinal surgery, spinal deformity, herniated disc, infection, fracture, myelopathy or malignancy, whiplash injury, systemic or neuromuscular disease, cognitive impairment) evaluated by medical history and diagnostics for images
* have previously undergone cognitive-behavioral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Neck Disability Index at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  Neck Disability Index, a self-administered 10-item questionnaire concerning neck pain disability, rates the intensity of pain and its disabling effects on typical daily activities. The score, expressed as a percentage, ranges from 0 (no disability) to 100 (maximum disability). Investigators used the Italian version which proved to be reliable and valid
Change from Baseline Tampa Scale of Kinesiophobia at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  Tampa Scale of Kinesiophobia is a self-report questionnaire that assesses pain beliefs and pain-related fear of movement/reinjury in subjects with musculoskeletal complaints. the 13-item Italian version ranges from 13 (best health status) to 52 (worst health status).
Change from Baseline Pain Catastrophizing Scale at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  Pain Catastrophizing Scale assesses catastrophizing in subjects with musculoskeletal complaints, and consists of a 13-item self-report questionnaire. The total score ranges from 0 to 52 with 52 indicating the worst health status.
  Investigators used the Italian version which proved to be reliable and valid.
Change from Baseline Numerical Rating Scale at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  Numerical Rating Scale assesses pain intensity using an 11-pointnumerical rating scale ranging from 0 (no pain) to10 (the worst imaginable pain).
Change from Baseline Short-Form Health Survey Questionnaire at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  Quality of life is assessed using the Italian version of the self-report Short-Form Health Survey with its eight domain scores ranging from 0 (the worst perceived quality of life) to 100 (the best perceived quality of life).
Change from Baseline Global Perceived Effect at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  Global Perceived Effect is a self-administered measure of treatment satisfaction consisting of a five-level Likert scale (1=helped a lot, 2=helped, 3=helped only a little, 4=did not help, 5=made things worse).

SECONDARY OUTCOMES:
Change from Baseline Work Ability Index at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  The Work Ability Index is an instrument used in occupational health care and research to assess work ability of workers exploring different dimensions; WAI is scored by summing the points received for each item: the best possible rating on the index is 49 points and the worst is 7 points.
Change from Baseline of Anamnestic survey of the upper limbs and spine's pathologies at 10 weeks and 12 months | Questionnaires will be administered before treatment, ten weeks after (post-treatment) and 12 months after the end of treatment (follow-up).
  Anamnestic and clinical evaluation of the pathologies affecting the upper limbs and spine, over the last 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Monticone, MD, PhD, Principal Investigator — Dept. Medical Sciences and Public Health, University of Cagliari, Cagliari, Italy
Locations (1):
- University of Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monticone M, Simone Vullo S, Lecca LI, Meloni F, Portoghese I, Campagna M. Effectiveness of multimodal exercises integrated with cognitive-behavioral therapy in working patients with chronic neck pain: protocol of a randomized controlled trial with 1-year follow-up. Trials. 2022 May 21;23(1):425. doi: 10.1186/s13063-022-06340-7. PMID 35597965

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04768790/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04768790/ICF_001.pdf